CLINICAL TRIAL: NCT00180050
Title: Efficacy and Safety of Budesonide for Treatment of Lymphocytic Colitis
Brief Title: Budesonide Treatment for Lymphocytic Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Dr. Falk Pharma GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BLYCK
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Microscopic Colitis
Keywords: lymphocytic colitis; microscopic colitis; budesonide
MeSH Terms: conditions — Colitis, Microscopic; Colitis, Lymphocytic | interventions — Budesonide

INTERVENTIONS:
Drug: Budesonide

SUMMARY:
The purpose of this study is to determine whether orale budesonide is effective in the treatment of lymphocytic colitis

DETAILED DESCRIPTION:
The purpose of this study is to determine whether orale budesonide is effective in the treatment of lymphocytic colitis

ELIGIBILITY:
Inclusion Criteria:

* lymphocytic colitis
* diarrhea
* effective contraception
* written informed consent

Exclusion Criteria:

* other forms if IBD
* celiac disease
* infectious colitis
* history of colonic surgery
* use of budesonide, 5-ASA, steroids within th previous 4 weeks
* pregnancy, lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2002-01; Primary Completion 2006-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in clinical remission after 6 weeks

SECONDARY OUTCOMES:
safety
quality of life
histological improvement

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Miehlke, Prof., Principal Investigator — Medical Department I, Technical University Hospital, Dresden, Germany
Locations (1):
- Medical Department I, Technical University Hospital, Dresden, Germany